CLINICAL TRIAL: NCT06814119
Title: A Clinical Study to Evaluate the Effect of Renal Impairment on the Single-Dose Pharmacokinetics of MK-1084
Brief Title: A Clinical Study of MK-1084 in Participants With Renal Impairment (MK-1084-010)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1084-010; MK-1084-010 (Other: MSD)
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Healthy; Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Panel A: Severe RI (Experimental): Participants with severe RI will be administered a single oral dose of MK-1084 on Day 1 under fasting conditions.
  Interventions: Drug: MK-1084
- Panel B: Moderate RI (Experimental): Participants with moderate RI will be administered a single oral dose of MK-1084 on Day 1 under fasting conditions.
  Interventions: Drug: MK-1084
- Panel C: Healthy (Experimental): Healthy participants will be administered a single oral dose of MK-1084 on Day 1 under fasting conditions.
  Interventions: Drug: MK-1084

INTERVENTIONS:
Drug: MK-1084 — Oral tablet

SUMMARY:
The goal of this study is to learn what happens to MK-1084 levels in a person's body over time. Researchers will measure what happens to MK-1084 levels in the body when it is given to people with moderate or severe renal impairment (RI) (meaning the kidneys do not work properly) as compared to people who are in good health. Researchers also want to learn about the safety of MK-1084 when it is given to people with RI and if people with RI can tolerate it.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

All participants:

- Has a BMI ≥18.0 and ≤40.0 kg/m^2

Participants with severe or moderate RI:

* With the exception of RI, is sufficiently healthy for study participation
* Has stable renal function with no clinically significant change in renal status at least 29 days prior to dosing and is not currently or has not been previously on dialysis for at least 1 year

Participants with normal renal function:

- Is medically healthy

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

All participants:

* Has a history of cancer (malignancy)
* Has positive results for human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C virus
* Has had major surgery and/or donated or lost significant volume of blood within 56 days prior to dosing

Participants with severe or moderate RI:

* Has a history or presence of renal artery stenosis
* Has a renal transplant or nephrectomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-11-21 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC0-inf) of MK-1084 | At designated timepoints (up to approximately 2 days postdose)
  Blood samples will be collected to determine the AUC0-inf of MK-1084.
Area Under the Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-last) of MK-1084 | At designated timepoints (up to approximately 2 days postdose)
  Blood samples will be collected to determine the AUC0-last of MK-1084.
Area Under the Concentration-Time Curve from Time 0 to 24 Hours (AUC0-24) of MK-1084 | At designated timepoints (up to 24 hours postdose)
  Blood samples will be collected to determine the AUC0-24 of MK-1084.
Plasma Concentration of MK-1084 at 24 Hours Postdose (C24) | At designated timepoints (up to 24 hours postdose)
  Blood samples will be collected to determine the C24 of MK-1084.
Maximum Plasma Concentration (Cmax) of MK-1084 | At designated timepoints (up to approximately 2 days postdose)
  Blood samples will be collected to determine the Cmax of MK-1084.
Time to Maximum Plasma Concentration (Tmax) of MK-1084 | At designated timepoints (up to approximately 2 days postdose)
  Blood samples will be collected to determine the Tmax of MK-1084.
Apparent Terminal Half-life (t1/2) of MK-1084 | At designated timepoints (up to approximately 2 days postdose)
  Blood samples will be collected to determine the t1/2 of MK-1084.
Apparent Clearance (CL/F) of MK-1084 | At designated timepoints (up to approximately 2 days postdose)
  Blood samples will be collected to determine the CL/F of MK-1084.
Apparent Volume of Distribution During Terminal Phase (Vz/F) of MK-1084 | At designated timepoints (up to approximately 2 days postdose)
  Blood samples will be collected to determine the Vz/F of MK-1084.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event | Up to approximately 2 weeks
  An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug. The number of participants who experience an adverse event will be reported.
Number of Participants Who Discontinue From the Study Due to an Adverse Event | Up to approximately 2 weeks
  An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug. The number of participants who discontinue from the study due to an adverse event will be reported.
Total Amount of MK-1084 Excreted Unchanged in Urine (Ae) | At designated timepoints (up to approximately 1 day postdose)
  Urine samples will be collected to determine the Ae of MK-1084.
Total Amount of MK-1084 Excreted Unchanged in Urine From 0 to 24 Hours (Ae0-24) | At designated timepoints (up to 24 hours postdose)
  Urine samples will be collected to determine the Ae0-24 of MK-1084.
Fraction of MK-1084 Excreted Unchanged in Urine (fe) | At designated timepoints (up to approximately 1 day postdose)
  Urine samples will be collected to determine the fe of MK-1084.
Renal Clearance (CLr) of MK-1084 | At designated timepoints (up to approximately 1 day postdose)
  Urine samples will be collected to determine the CLr of MK-1084.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Orlando Clinical Research Center ( Site 0002), Orlando, Florida
  - Research by Design ( Site 0001), Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/